CLINICAL TRIAL: NCT01694550
Title: Corrected QT Interval in Patients With Pacemaker Dependency (QT-TENDENCY-Study)
Brief Title: QT Interval in Patients With Pacemaker Dependency
Acronym: QT-TENDENCY
Status: Completed | Type: Observational
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Dr. Samir Said, Dr. med., University of Magdeburg
Other Study IDs: OVGU-Kar-011
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: High Degree AV-block; Left Bundle Branch Block
Keywords: pacemaker; ICD / CRTD; corrected QT-interval
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimen are necessary for the study and this issue is irrelevant.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pacemaker mode programming: High grade AV-block

SUMMARY:
The aim of this study is to examine a correction term for an adapted QT interval during ventricular pacing (right, left and biventricular pacing) to obtain valid formulae correcting for the QT intervals in various pacing conditions.

DETAILED DESCRIPTION:
This investigation aims at determining a possibility to assess the usefulness of various formulae that correct for the different effects of various pacing modes on the QT interval. More specifically, the hypothesis will be tested that applying adequate correction will preserve the predictive power of the QT-interval regarding proarrhythmia in various cardiac pathologies and therapies.

ELIGIBILITY:
Inclusion Criteria:

* caucasian race
* implanted cardioverter/defibrillator or pacemaker
* negative pregnancy test for women of child bearing potential
* stable function of the implanted device
* stable medical therapy relating to the underlying disease
* stable medical therapy of antiarrhythmic drugs and other QT-time changing drugs
* no instability of rhythm
* x-ray of thorax during device implantation in two levels (ap and ll axis)
* written informed consent

Exclusion Criteria:

* coronary heart disease and angina pectoris symptoms
* patient with acute myocardial infarction or CABG while the last 4 weeks
* patient with tachycardia and a rest frequency >80 bpm
* patient with severe pulmonary disease
* patient with anaemia
* patient with acute infections
* patient with severe kidney or liver disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll 180 patients after an implantation of cardioverter/defibrillator or pacemaker based on a standard guideline indication. The point of enrolment for all patients is the time at which the patient signs and dates the ICF during the hospital stay in the context of implantation.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Corrected QT Interval in Patients With Pacemaker Dependency | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Samir Said, Dr., Principal Investigator — Magdeburg University
Locations (1):
- Magdeburg University, Internal Medicine/Cardiology, Angiology and Pneumologie, Magdeburg, Germany